CLINICAL TRIAL: NCT00583973
Title: The Effect of Parenteral Iron Therapy on the Systemic Inflammatory Response and Oxidative Stress in Chronic Hemodialysis Patients
Brief Title: Effect of Parenteral Iron Therapy on Inflammatory Response and Oxidative Stress Chronic Hemodialysis
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200614206
Record Dates: First submitted 2007-12-22; First posted 2008-01-02 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Hemodialysis; Chronic Kidney Disease; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Chronic hemodialysis patients

SUMMARY:
Parenteral iron therapy is now commonly administered to dialysis patients with the majority of patients receiving this therapy as part of the treatment for their anemia. Although intravenous iron has improved clinical response to recombinant erythropoietin, there is a concern that iron therapy may have deleterious effects in Chronic Kidney Disease (CKD) patients. Iron can damage tissues by catalyzing the conversion of hydrogen peroxide to free-radical ions that attack cellular proteins, DNA and membranes as part of oxidative stress. Numerous in vitro studies have shown tissue toxicity from iron and increased infectious potential. Oxidative stress can also lead to activation of the systemic inflammatory response with the release of a number of key cytokines and growth factors. There is now a link between inflammation, oxidative stress and acceleration of vascular disease in both patients with normal as well as reduced renal function. In a study comparing normal versus low hematocrit levels in hemodialysis patients, mortality was higher in the normal hematocrit group. The major difference between the two groups has been attributed to the fact that patients in the normal hematocrit group received significantly more iron than the patients with low hematocrit. There was a 2.4 fold greater mortality rate in patients receiving parenteral iron.

The effect of parenteral iron administration on activation of the systemic inflammatory response in hemodialysis patients has not been evaluated. The purpose of this study is to measure a number of key cytokines, inflammatory and oxidative stress markers in hemodialysis patients receiving iron repletion therapy as part of their standard care.

DETAILED DESCRIPTION:
Study Design

Patients who have been prescribed iron repletion therapy (100 mg IV every dialysis treatment for ten treatments) by their primary nephrologist will be recruited for the study. Baseline blood samples will be obtained before and after each dialysis treatment for two dialysis treatments prior to the administration of iron. On the day of dialysis that iron therapy is started, blood samples will be obtained before and after the dialysis treatment via the patient's vascular access. This procedure will be repeated each dialysis treatment for the ten sessions during which the patient is receiving intravenous iron. Subsequently, pre-dialysis blood samples will be obtained every week for four weeks after the administration of intravenous iron has been completed

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients age 18 or greater who are prescribed parenteral iron by their primary nephrologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hemodialysis patients--stage V CKD
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burl R Don, MD, Principal Investigator — University of California, Davis
Locations (1):
- Dialysis Clinics Inc, Sacramento, California, United States